CLINICAL TRIAL: NCT06459583
Title: Evaluation of Self-Mediated Alternatives for Risk Testing Education and Return of Results
Acronym: eSMARTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Banner Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: API-0001; R01AG058468 (NIH)
Record Dates: First submitted 2024-05-23; First posted 2024-06-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
Keywords: APOE
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth platform (Experimental): The eHealth platform consists of the self-directed web-portal (ADWebPortal) and chatbot (ADChatbot) to receive their Alzheimer's-related test results. Participants randomized to this arm can switch between the two or schedule a virtual appointment with a healthcare provider.
  Interventions: Other: eHealth Platform
- Videoconference telehealth (Active Comparator): The videoconference telehealth platform consists of remote visit(s) with a healthcare provider to receive their Alzheimer's-related test results.
  Interventions: Other: Videoconference Telehealth Platform

INTERVENTIONS:
Other: eHealth Platform — The eHealth Platform consists of the ADWebPortal and ADChatbot for receiving Alzheimer's-related test results
  Arms: eHealth platform
Other: Videoconference Telehealth Platform — Participants will have a video telehealth visit with a healthcare provider to receive Alzheimer's-related test results
  Arms: Videoconference telehealth

SUMMARY:
This randomized non-inferiority study will evaluate self-directed scalable electronic health platform (eHealth) methods for communicating Alzheimer's gene and biomarker results compared to videoconference telehealth disclosure with healthcare providers, as well as characterize the impacts of learning this information on the participant.

DETAILED DESCRIPTION:
This is a randomized trial to evaluate self-directed scalable eHealth methods for communicating Alzheimer's gene and biomarker results, as well as characterize the clinical impacts of learning this information on the participant. All participants in the study will be randomized to receive their Alzheimer's gene and biomarker results either via person-mediated telehealth videoconference visit with a healthcare provider or by eHealth platform. A permuted block design will be used for randomization, and we will stratify by sex and apolipoprotein E (APOE) genotype.

Participants randomized to the eHealth arm will be offered either the ADWebPortal or ADChatbot but can switch between platforms or schedule a virtual appointment to speak with a healthcare provider at any point. Use of the pre-disclosure education platforms will be tracked. A HIPAA compliant telehealth application will be used for the person-mediated telehealth videoconference visits and sessions will be recorded.

Potential participants will be identified from the GeneMatch program. Study management and participation will be decentralized. Confirmation of eligibility and consent of potential participants will be completed remotely by a decentralized study team. Procedures requiring physical attendance (e.g., blood draw) will be completed remotely using mobile health services.

ELIGIBILITY:
Inclusion Criteria:

* Access to the internet and an internet-enabled device.
* Participant is able to provide informed consent as shown by correctly answering questions administered by the study coordinator during the electronic consenting process that assess understanding of consent form content.
* Participant is willing and has the ability to fully comply with study procedures defined in this protocol.
* Written and spoken fluency in the English.
* Participant agrees to undergo a blood draw for collection of a blood sample for future testing and repository storage.

Exclusion Criteria:

* Participant reports prior knowledge of APOE genotype.
* Lack of psychological readiness to receive AD gene and biomarker information as indicated by:

  1. obtaining a score of 10 or greater on the Patient Health Questionnaire - 9 (PHQ-9) AND/OR
  2. responding yes on any of the suicidal ideation questions extracted from the abbreviated Columbia Suicide Severity Scale (C-SSRS) or AD Specific Suicidality Questions.
* Presence of current major psychiatric illness, e.g., psychosis, bipolar disorder, PTSD
* Communication difficulties such as:

  1. Uncorrected or uncompensated hearing and/or vision impairment.
  2. Uncorrected or uncompensated speech defects.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 681 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-11-07 (Actual); Study Completion 2025-11-07 (Actual)

PRIMARY OUTCOMES:
Anxiety as measured by the PROMIS Anxiety scale | T2 minus T1 change scores (6-weeks post disclosure minus 0-7 days post disclosure)
  Anxiety scale
Knowledge of Genetic Disease as measured by an 8-item scale adapted from the Cancer Genetics Knowledge Scale and ClinSeq Knowledge Scale | T2 minus T1 change scores (6-weeks post disclosure minus 0-7 days post disclosure)
  Knowledge of Genetic Disease scale
Disease-specific distress as measured by an 8-item scale adapted from the Impact of Events Scale | T2 minus T1 change scores (6-weeks post disclosure minus 0-7 days post disclosure)
  Disease-specific distress scale

SECONDARY OUTCOMES:
Depression as measured by the Patient Health Questionnaire - 9 (PHQ-9) | 0-7 days, 6 weeks, 6 months
  Depression scale
Psychological wellbeing as measured by a 14-item scale adapted from the Psychological Wellbeing Scale | 6 months
  Psychological wellbeing scale
Perceived risk of Alzheimer's as measured by a scale adapted from the REVEAL Study | 0-7 days, 6 weeks, 6 months
  Perceived risk of Alzheimer's scale
Impact of disclosure as measured by the 16-item IGT-AD scale | 0-7 days, 6 weeks, 6 months
  Impact of genetic testing for Alzheimer's disease (IGT-AD) scale
Subjective cognitive concerns as measured by the 14-item Cognitive Function Instrument | 6 months
  Subjective cognitive concerns scale
Stigma as measured by the 6-item Stigma Impact Scale | 0-7 days, 6 weeks, 6 months
  Stigma scale

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Langbaum, PhD, Principal Investigator — Banner Alzheimer's Institute
Locations (2):
- United States (2):
  - Accellacare Clinical Research Site 02, Mt. Pleasant, South Carolina
  - Accellacare Clinical Research Site 01, Bristol, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Trial dataset and biological samples will be shared with qualified investigators
Supporting Information: Study Protocol
Time Frame: Data will be shared within 12 months after study completion

REFERENCES:
- [Background] Erickson CM, Langlois CM, Wood EM, Mim R, Howe S, Ofidis D, Egleston BL, Harkins K, Largent EA, Roberts JS, Reiman EM, Denkinger M, Ashton NJ, Karlawish J, Bradbury AR, Langbaum JB. Evaluation of self-mediated alternatives for risk testing education and return of results (eSMARTER) study: A randomized study of methods for returning APOE and pTau-217 results. Alzheimers Dement (N Y). 2025 Nov 16;11(4):e70177. doi: 10.1002/trc2.70177. eCollection 2025 Oct-Dec. PMID 41250770